CLINICAL TRIAL: NCT04796701
Title: Effect of a Transitional Care Intervention From Hospital to Home on Readmissions Among Older Medical Patients: a Quasi-experimental Study.
Brief Title: Effect of a Transitional Care Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FH2017-2019
Record Dates: First submitted 2021-02-24; First posted 2021-03-15 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-02

CONDITIONS: Frailty
Keywords: readmission; transitional care; discharge; older medical patients
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled trial
Masking Description: Intervention group: living in three predefined municipality Control group: living in one predefined municipality
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follow Home Intervention (Experimental): If possible, all included participants are physically followed home by a hospital-based project worker on the day of discharge. During the visit, the focus is on: basic human needs, medication review reconciliation, and a comprehensive geriatric assessment. Problems, challenges and concerns are discussed. Finally, a conference for the following working day is arranged either as a physical visit or a video conference. The patient, relatives, community-based nurse and project worker are invited to participate and health status and challenges are discussed They are recommended to contact the project worker about health and practical issues up to 7 days after discharge where the intervention ends. Subsequently, the responsibility for treatment and care is assigned to the GP and home healthcare provider.
  Interventions: Other: Follow-Home-intervention
- Control (No Intervention): On the day of discharge, the hospital-based nurse digitally sends a summary of the hospital stay and a treatment and care plan to the community-based nurse. If needed, the hospital-based nurse contacts the community-based nurse by phone as a supplement to the plan. Finally, a discharge letter conducted by the hospital-based doctor is digitally sent to the GP

INTERVENTIONS:
Other: Follow-Home-intervention — x
  Arms: Follow Home Intervention

SUMMARY:
The objective of this study is to evaluate the effect of a transitional care intervention on readmissions among older medical patients.

The proportion of older people is rapidly growing. These changes represent a challenge for healthcare systems. 20% of all hospital admitted patients ≥ 65 years are readmitted within the first 30 days after discharge. Prior transitional care research has mainly focused on either hospital-based or community-based interventions with no or little intervention elements in both settings. The results show different effects on readmission rates. This calls for new research on trans-sectorial interventions with both pre- and post-discharge elements.

DETAILED DESCRIPTION:
Design:

Non-randomized controlled trial.

Participants For eligibility criteria - see elsewhere. Intervention group • Patients living in Odder, Skanderborg or Hedensted municipality

Control group

• Patients living in Horsens municipality

Follow-Home Intervention

The intervention group receives following intervention:

If possible, all included participants are physically followed home by a hospital-based project worker on the day of discharge. During the visit, the focus is on: basic human needs, medication review reconciliation, and a comprehensive geriatric assessment. Problems, challenges and concerns are discussed. Finally, a conference for the following working day is arranged either as a physical visit or a video conference. The patient, relatives, community-based nurse and project worker are invited to participate and health status and challenges are discussed They are recommended to contact the project worker about health and practical issues up to 7 days after discharge where the intervention ends. Subsequently, the responsibility for treatment and care is assigned to the GP and home healthcare provider.

Usual care

Patients in the control group recieves the following usual discharge procedure:

On the day of discharge, the hospital-based nurse digitally sends a summery of the hospital stay and a treatment and care plan to the community-based nurse. If needed, the hospital-based nurse contacts the community-based nurse by phone as a supplement to the plan. Finally, a discharge letter conducted by the hospital-based doctor is digitally sent to the GP.

Method:

Inclusion of participants is consecutive. Inclusion period was between 01/02/17 to 31/12/19. In total, approximately 1200 patients were included .

Data collection Outcome data will be retrieved from CROSS-TRACKS database at 30 days after discharge from index admission.

Analysis

Intervention and Control group will be matched on 3 variables on individual level:

* CCI
* Index admission period: +/- 3-4 weeks
* Sex

All readmissions are included in the analysis (not only first time readmissions). That means that one patient can be included several times.

Logistic regression adjusted for possible confounders will be used when analysing the outcomes. Confounders are chosen through a study specific DAG.

Sub-group analysis will be conducted according to:

* Age
* Sex
* Housing
* Civil status
* Social status
* Length of hospital stay in index admission
* Comorbidity
* Diagnosis
* Ect.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥75 years
* Living in the municipalities of Odder, Skanderborg, Hedensted or Horsens
* Admitted for ≥48 hours
* Discharged from Medical Ward 1 (MSA1) at Horsens Regional Hospital (HRH)

Exclusion Criteria:

* Terminally ill patients
* Patients with cerebrovascular events
* Readmitted to another hospital
* Not able to speak and understand Danish

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1266 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Readmission | Readmission will be assessed at 30 days after hospital discharge in both intervention and control group
  Unplanned all-cause readmission

SECONDARY OUTCOMES:
Mortality | Mortality will be assessed at 30 days after hospital discharge in both intervention and control group
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Merete Gregersen, PHD, Study Chair — Aarhus University Hospital
Locations (1):
- Horsens Regional Hospital, Horsens, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rasmussen LF, Barat I, Riis AH, Gregersen M, Grode L. Effects of a transitional care intervention on readmission among older medical inpatients: a quasi-experimental study. Eur Geriatr Med. 2023 Feb;14(1):131-144. doi: 10.1007/s41999-022-00730-5. Epub 2022 Dec 23. PMID 36564644